CLINICAL TRIAL: NCT01967290
Title: Phase II Study of the Impact of the SWORD Device on Rehabilitation Tasks Performance in the Early Post Stroke Period
Brief Title: Stroke Wearable Operative Rehabilitation Device Impact Trial
Acronym: SWORD-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar de Entre o Douro e Vouga (Other)
Responsible Party: Principal Investigator, Vítor Tedim Cruz, MD, Centro Hospitalar de Entre o Douro e Vouga
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PTDC/SAU-NEU/102075/2008_SWORD
Record Dates: First submitted 2013-10-18; First posted 2013-10-22 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Ischemic Stroke; Upper Extremity Hemiparesis
Keywords: stroke; motor deficits; motor rehabilitation; neurorehabilitation; medical devices; wearable devices; e-health systems
MeSH Terms: conditions — Ischemic Stroke; Stroke; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hand-to-mouth task - vibratory feedback (Experimental): Hand-to-mouth task under vibratory feedback and 3D movement analysis. The SWORD device is in place over the patient arm, performs continuous 3D movement analysis and provides vibratory feedback according to quality performance settings established by the clinician after patient assessment. If movement is of lower amplitude or slower than prescribed a vibratory stimulus is delivered at the wrist of the patient. The intervention is repeated on the hemiparetic and normal sides and the duration of the task is defined according to the patient cardiovascular status.
  Interventions: Device: Vibratory feedback and 3D movement analysis
- Hand-to-mouth task - no vibratory feedback (Active Comparator): Hand-to-mouth task in the same conditions as the experimental arm but without vibratory feedback, only 3D movement analysis. The SWORD device is in place over the patient arm, performs continuous 3D movement analysis but does not provides vibratory feedback according to quality performance settings established by the clinician after patient assessment. If movement is of lower amplitude or slower than prescribed NO vibratory stimulus is delivered at the wrist of the patient. The intervention is repeated on the hemiparetic and normal sides and the duration of the task is defined according to the patient cardiovascular status.
  Interventions: Device: Only 3D movement analysis

INTERVENTIONS:
Device: Vibratory feedback and 3D movement analysis — Hand-to-mouth task performed under vibratory feedback combined with 3D continuous movement analysis.
  Other Names: Propriocetive actuation; Vibratory stimulation; SWORD; Stroke Wearable Operative Rehabilitation Device
  Arms: Hand-to-mouth task - vibratory feedback
Device: Only 3D movement analysis — Hand-to-mouth task performed under 3D continuous movement analysis only
  Other Names: 3D movement quantification; 3D movement characterization; SWORD; Stroke Wearable Operative Rehabilitation Device
  Arms: Hand-to-mouth task - no vibratory feedback

SUMMARY:
The objective of this study is to determine the impact of vibratory feedback on the quality and intensity of a common motor rehabilitation task of the upper-arm (hand-to-mouth) in stroke patients. For that purpose the investigators use the SWORD system that combines 3D motion quantification wearable sensors and a vibratory module.

The investigators hypothesize that vibratory stimuli during a motor rehabilitation task increase significantly the number of correct movements performed per unit of time.

The design of the study is a cross-over randomized clinical trial. With the SWORD system in place each patient will perform the hand-to-mouth task twice (with vibratory feedback and without it), the order being random. The number of correct movements and other motor outcomes will be assessed continuously under both conditions.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old at stroke onset, with no superior age limit;
* Medical diagnosis of acute ischemic stroke;
* First ever stroke;
* Previously independent, defined as having a modified Rankin scale (mRS) of 0-1;
* Clinical and CT or MRI compatible with a medial cerebral artery ischemic lesion;
* Confirmed motor deficit on the upper limb but not plegia (able to actively extend wrist, thumb, and at least 2 other digits >10°), defined as a score between 0 and 2 on items 5a or 5b of the National Institute of Health Stroke Scale;
* Inpatients, within no more than 4 weeks after stroke onset;
* Medically stable, no intravenous medication and already able to sit for more than one hour comfortably;
* Favourable opinion of the attending stroke physician;
* Patient and caregiver understand the purpose of the study and provided written informed consent.

Exclusion Criteria:

* No detectable motor deficits at baseline assessment by the neurologist;
* Severe aphasia;
* Dementia (any stage);
* Other cognitive or psychiatric comorbidity that impairs communication or compliance with the tasks;
* Severe respiratory or cardiac condition incompatible with more than one minute of continuous mild exercise (e.g. combing hair) in a sitting position;
* Pain that limits upper limb movement either on the normal or affected side;
* Upper limb amputation or severe deformity either on the normal or affected side;
* Fixed articular limitations of upper limb either on the normal or affected side;
* Enrollment in other trial in the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of correct movements | At the end of each hand-to-mouth task.
  Number of correct movements performed within the duration of each hand-to-mouth task.

SECONDARY OUTCOMES:
Total number of movements | At the end of each hand-to-mouth task.
  Total number of correct and incorrect movements performed within the duration of each hand-to-mouth task.
Range of motion in degrees | At the end of each hand-to-mouth task.
  Average, standard deviation and variance of the range of motion, measured in degrees, of all the correct movements performed during the duration of each hand-to-mouth task.
Time between correct movements in seconds | At the end of each hand-to-mouth task.
  Average, standard deviation and variance of the time between correct movements, measured in seconds, of all the correct movements performed during the duration of each hand-to-mouth task.
Cumulative amplitude of correct movements in degrees | At the end of each hand-to-mouth task
  Sum of the amplitudes of all correct movements performed within the duration of each hand-to-mouth task.
Cumulative amplitude of all movements performed in degrees | At the end of each hand-to-mouth task.
  Sum of the amplitudes of all correct and incorrect movements performed within the duration of each hand-to-mouth task.
Number of pause events during the task | At the end of each hand-to-mouth task
  Number of episodes during the execution of each hand-to-mouth task where the patient stopped doing movements and/or the time between correct movements exceeded the mean plus one standard deviation measured within the same hand-to-mouth task.
Fatigue | At the end of each hand-to-mouth task.
  Assessment of fatigue by the patient through an analogic scale from 0 (no fatigue) to 4 (interruption due to fatigue).
Pain | At the end of each hand-to-mouth task.
  Assessment of pain by the patient through an analogic scale from 0 (no pain) to 4 (interruption due to pain).
Number and type of other distresses | At the end of each hand-to-mouth task.
  Recording and description of any kind of discomfort reported by the patient or detected through vital parameter and arterial oxygen saturation monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Vítor T. Cruz, MD, Principal Investigator — Centro Hospitalar de Entre o Douro e Vouga; Paula Coutinho, PhD, Study Chair — IBMC - University of Oporto
Locations (3):
- Portugal (3):
  - Rehabilitation Department, Centro Hospitalar do Alto Ave, EPE, Guimarães
  - Neurology Department, CHEDV, Santa Maria da Feira
  - Rehabilitation Department, CHEDV, Santa Maria da Feira

REFERENCES:
- [Background] Bento VF, Cruz VT, Ribeiro DD, Cunha JP. The vibratory stimulus as a neurorehabilitation tool for stroke patients: proof of concept and tolerability test. NeuroRehabilitation. 2012;30(4):287-93. doi: 10.3233/NRE-2012-0757. PMID 22672942
- [Background] Bento VF, Cruz VT, Ribeiro DD, Cunha JP. Towards a movement quantification system capable of automatic evaluation of upper limb motor function after neurological injury. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:5456-60. doi: 10.1109/IEMBS.2011.6091392. PMID 22255572
- [Background] Bento VF, Cruz VT, Ribeiro DD, Colunas MM, Cunha JP. The SWORD tele-rehabilitation system. Stud Health Technol Inform. 2012;177:76-81. PMID 22942034
- [Background] Bento VF, Cruz VT, Ribeiro DD, Branco C, Coutinho P. The potential of motion quantification systems in the automatic evaluation of motor function after stroke. Int J Stroke. 2013 Aug;8(6):E37. doi: 10.1111/ijs.12111. No abstract available. PMID 23879761
- [Derived] Cruz VT, Bento V, Ruano L, Ribeiro DD, Fontao L, Mateus C, Barreto R, Colunas M, Alves A, Cruz B, Branco C, Rocha NP, Coutinho P. Motor task performance under vibratory feedback early poststroke: single center, randomized, cross-over, controlled clinical trial. Sci Rep. 2014 Jul 11;4:5670. doi: 10.1038/srep05670. PMID 25011667